CLINICAL TRIAL: NCT00857545
Title: A Phase II Randomized, Double-Blind Trial of a Polyvalent Vaccine-KLH Conjugate (NSC 748933 ) + OPT-821 Versus OPT-821 in Patients With Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer Who Are in Second or Third Complete Remission
Brief Title: OPT-821 With or Without Vaccine Therapy in Treating Patients With Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Peritoneal Cancer in Second or Third Complete Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GOG-0255; NCI-2009-01176 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000636384; GOG-0255 (Other: NRG Oncology); GOG-0255 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2016-12

CONDITIONS: Stage IA Fallopian Tube Cancer; Stage IA Ovarian Cancer; Stage IB Fallopian Tube Cancer; Stage IB Ovarian Cancer; Stage IC Fallopian Tube Cancer; Stage IC Ovarian Cancer; Stage IIA Fallopian Tube Cancer; Stage IIA Ovarian Cancer; Stage IIB Fallopian Tube Cancer; Stage IIB Ovarian Cancer; Stage IIC Fallopian Tube Cancer; Stage IIC Ovarian Cancer; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (vaccine therapy and adjuvant) (Experimental): Patients receive polyvalent antigen-KLH conjugate vaccine and immunological adjuvant OPT-821 subcutaneously (SC) once in weeks 1, 2, 3, 7, 11, 23, 35, 47, 59, 71, and 83 in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Polyvalent Antigen-KLH Conjugate Vaccine; Biological: Saponin-based Immunoadjuvant OBI-821
- Arm II (adjuvant) (Experimental): Patients receive immunological adjuvant OPT-821 SC as in arm I.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Saponin-based Immunoadjuvant OBI-821

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Polyvalent Antigen-KLH Conjugate Vaccine — Given SC
  Arms: Arm I (vaccine therapy and adjuvant)
Biological: Saponin-based Immunoadjuvant OBI-821 — Given SC
  Other Names: OBI-821; OPT-821

SUMMARY:
This randomized phase II trial studies OPT-821 and vaccine therapy to see how well they work compared with OPT-821 alone in treating patients with ovarian epithelial cancer, fallopian tube cancer, or peritoneal cancer that has decreased or disappeared, but the cancer may still be in the body. Biological therapies, such as OPT-821, may stimulate the immune system in different ways and stop tumor cells from growing. Vaccines may help the body build an effective immune response to kill tumor cells. It is not yet known whether OPT-821 is more effective with or without vaccine therapy in treating patients with ovarian epithelial cancer, fallopian tube cancer, or peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if a polyvalent vaccine (including GM2-keyhole limpet hemocyanin [KLH], Globo-H-KLH, Tn-mucin 1 [MUC1]-32mer-KLH, and Thompson Friedreich antigen [TF]-KLH plus OPT-821) decreases the hazard of progression or death compared to a vaccine containing OPT-821 alone in women with epithelial ovarian, fallopian tube, or peritoneal cancer in second or third complete clinical remission.

SECONDARY OBJECTIVES:

I. To compare the treatment arms with respect to the incidence of toxicities. II. To determine if the polyvalent vaccine decreases the hazard of death compared to a vaccine containing OPT-821 alone in women with epithelial ovarian, fallopian tube, or peritoneal cancer in second or third complete clinical remission.

TERTIARY OBJECTIVES:

I. To evaluate the immune response (by enzyme linked immunosorbent assay [ELISA]) in participants, in order to determine if the outcome correlates with antigen-specific immune titers.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive polyvalent antigen-KLH conjugate vaccine and immunological adjuvant OPT-821 subcutaneously (SC) once in weeks 1, 2, 3, 7, 11, 23, 35, 47, 59, 71, and 83 in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive immunological adjuvant OPT-821 SC as in Arm I.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented epithelial carcinoma arising in the ovary, fallopian tube, or peritoneum, of any stage or grade at diagnosis; all patients must have had cytoreductive surgery and chemotherapy with at least one platinum-based chemotherapy regimen as part of primary treatment
* Patients who recurred on or after initial therapy, and are now in a second or third complete clinical remission and who are within four months of their last treatment are eligible; complete clinical remission is defined as serum cancer antigen (CA)-125 within institutional normal limits, negative physical examination, and no definite evidence of disease by computed tomography (CT) of the abdomen and pelvis; lymph nodes and/or soft tissue abnormalities =< 1.0 cm are often present in the pelvis and will not be considered definite evidence of disease; eligibility is determined by anatomical imaging only (ie. magnetic resonance imaging [MRI] or CT); a positive positron emission tomography (PET) image (if performed) will not exclude a patient if other criteria are met and anatomical imaging is negative
* Absolute neutrophil count (ANC) greater than or equal to 1,000/mm^3, equivalent to Common Toxicity Criteria for Adverse Events (CTCAE version [v]4.0) grade 1
* Platelets greater than or equal to 100,000/mm^3
* Serum creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), CTCAE v4.0 grade 1
* Bilirubin less than or equal to 2.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT), serum glutamate pyruvate transaminse (SGPT) less than or equal to 2.5 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Patients must have a Gynecological Oncology Group (GOG) performance status of 0, 1, or 2
* Patients who have signed the informed consent document and signed the authorization permitting release of personal health information
* Patients of childbearing potential must have a negative serum pregnancy test prior to study entry and must be practicing an effective form of birth control; nursing mothers are excluded

Exclusion Criteria:

* With the exception of non-melanoma skin cancer, patients with other invasive malignancies who had (or have) any evidence of the other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy are excluded
* Patients whose circumstances at the time of entry onto the protocol would not permit completion of study or required follow up
* Patients who have an allergy to shellfish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2010-07; Primary Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, Principal Investigator — NRG Oncology
Locations (45):
- United States (45):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Saint Vincent Oncology Center, Indianapolis, Indiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Gynecologic Oncology of West Michigan PLLC, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - The Women's Institute for Gynecologic Cancer and Special Pelvic Surgery, Phillipsburg, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] O'Cearbhaill RE, Deng W, Chen LM, Lucci JA 3rd, Behbakht K, Spirtos NM, Muller CY, Benigno BB, Powell MA, Berry E, Tewari KS, Hanjani P, Lankes HA, Aghajanian C, Sabbatini PJ. A phase II randomized, double-blind trial of a polyvalent Vaccine-KLH conjugate (NSC 748933 IND# 14384) + OPT-821 versus OPT-821 in patients with epithelial ovarian, fallopian tube, or peritoneal cancer who are in second or third complete remission: An NRG Oncology/GOG study. Gynecol Oncol. 2019 Dec;155(3):393-399. doi: 10.1016/j.ygyno.2019.09.015. Epub 2019 Oct 22. PMID 31653510

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 7/26/2010 and closed to accrual on 2/4/2013.
Groups:
- Polyvalent Antigen-KLH+OPT-821 Vaccine: Polyvalent antigen-KLH + OPT-821 vaccine subcutaneously administered on weeks 1, 2, 3, 7, 11, 23, 35, 47, 59, 71 and 83 for a total of 11 vaccines until disease progression or adverse effects prohibit further treatment. 1 cycle = 1 vaccine
- Non-specific Immunity With OPT-821: Non-specific OPT-821 subcutaneously administered on weeks 1, 2, 3, 7, 11, 23, 35, 47, 59, 71 and 83 for a total of 11 vaccines until disease progression or adverse effects prohibit further treatment. 1 cycle = 1 vaccine
Period: Overall Study
Arm/Group | Polyvalent Antigen-KLH+OPT-821 Vaccine | Non-specific Immunity With OPT-821
Started | 86 | 85
Completed | 86 (Enrolled and randomized participants.) | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled and randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Polyvalent Antigen-KLH+OPT-821 Vaccine | Non-specific Immunity With OPT-821 | Total
Number analyzed (Participants) | 86 | 85 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.6) | 59.1 (9.1) | 60.2 (8.9)
Age, Customized [Count of Participants; unit: Participants]
  40-49 | 8 | 14 | 22
  50-59 | 29 | 31 | 60
  60-69 | 37 | 26 | 63
  70-79 | 10 | 14 | 24
  80-89 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 85 | 171
  Male | 0 | 0 | 0
Recurring and/or Persistent Disease [Count of Participants; unit: Participants] — Recurrent/persistent patients
  Participants | 86 | 85 | 171
Cell Type [Count of Participants; unit: Participants]
  Adenocarcinoma with Squam. Diff ' n | 0 | 1 | 1
  Adenocarcinoma, Unsp. | 3 | 1 | 4
  Adenosquamous | 2 | 0 | 2
  Clear Cell Carcinoma | 1 | 1 | 2
  Endometrioid Adenocarcinoma | 6 | 1 | 7
  Mixed Epithelial Carcinoma | 2 | 2 | 4
  Other Carcinoma | 2 | 0 | 2
  Serous Adenocarcinoma | 69 | 76 | 145
  Transitional Cell Carcinoma | 0 | 2 | 2
  Undifferentiated Carcinoma | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is the period of time from the date of randomization to the date of first clinical, biochemical, or radiological evidence of progression, death due to any cause or date of last contact, whichever occurs first. Progression is defined as increasing clinical, radiological or histological evidence of disease. Patients with progressing disease based on clinical or histologic basis (ie. biopsy) must also have CT scan of the abdomen and pelvis performed.
Time Frame: Every 3 month until 2 years from start of treatment, then every 6 months for 3 years; then annually if patient remains in remission.
Population: Enrolled and randomized participants. 95% two-sided confidence interval
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Polyvalent Antigen-KLH+OPT-821 Vaccine | Non-specific Immunity With OPT-821
Number analyzed (Participants) | 86 | 85
Months | 5.9 [5.4 to 7.7] | 6.5 [5.1 to 7.9]

2. Secondary Outcome: Incidence of Adverse Effects (Grade 3 or Higher) During Treatment Period
Description: Number of participants with a maximum grade of 3 or higher during treatment period. Adverse events are graded and categorized using CTCAE v4.0.
Time Frame: During treatment period and up to 30 days after stopping the study treatment; up to 83 weeks.
Population: Enrolled and randomized and treated Patients. Grade 3 or worse adverse events for gastrointestinal disorders were significantly associated with treatment arm at significant level of 0.05 by two-sided Fisher's exact test. The reporting arm 2 had higher proportion of patients with reported grade 3 or worse adverse events.
Measure: Number; unit: participants
Arm/Group | Polyvalent Antigen-KLH+OPT-821 Vaccine | Non-specific Immunity With OPT-821
Number analyzed (Participants) | 86 | 85
participants
  Leukopenia | 0 | 0
  Thrombocytopenia | 0 | 0
  Neutropenia | 1 | 1
  Anemia | 0 | 1
  Other Investigations | 1 | 0
  Eye disorders | 0 | 1
  Gastrointestinal Disorders | 2 | 10
  General disorders & administration site condition | 1 | 0
  Immune system disorders | 0 | 1
  Infections and infestations | 1 | 0
  Metabolism and nutrition disorders | 3 | 1
  Neoplasms benign, malignant & unspecified | 2 | 0
  Nervous System | 1 | 1
  Psychiatric disorders | 1 | 0
  Renal and urinary disorders | 1 | 0
  Vascular disorders | 0 | 2

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death due to any cause or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years of follow-up.
Population: Enrolled and randomized participants. The upper limit of the 95% confidence interval for OS median in arm 1 is not available because the data is not mature enough for estimation at the time of this report.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Polyvalent Antigen-KLH+OPT-821 Vaccine | Non-specific Immunity With OPT-821
Number analyzed (Participants) | 86 | 85
Months | 46.5 [36.4 to NA] — As of date of submission, data is not mature enough to evaluate median confidence interval. | 46.2 [29.6 to 50.5]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported.
Arm/Group | Polyvalent Antigen-KLH+OPT-821 Vaccine | Non-specific Immunity With OPT-821
Serious Adverse Events (participants affected / at risk) | 5/86 | 14/84
Other Adverse Events (participants affected / at risk) | 84/86 | 82/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Polyvalent Antigen-KLH+OPT-821 Vaccine (N=86) | Non-specific Immunity With OPT-821 (N=84)
Colonic Obstruction (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 5
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Ileal Obstruction (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Autoimmune Disorder (Immune system disorders) | 0 | 1
Skin Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Neoplasms Benign, Malignant And Unspecified (Incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Personality Change (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Polyvalent Antigen-KLH+OPT-821 Vaccine (N=86) | Non-specific Immunity With OPT-821 (N=84)
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 31 | 33
Palpitations (Cardiac disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 2
Hearing Impaired (Ear and labyrinth disorders) | 1 | 2
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 3 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Eye Disorders - Other (Eye disorders) | 0 | 1
Watering Eyes (Eye disorders) | 1 | 0
Scleral Disorder (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Blurred Vision (Eye disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 15 | 16
Diarrhea (Gastrointestinal disorders) | 6 | 5
Vomiting (Gastrointestinal disorders) | 5 | 10
Bloating (Gastrointestinal disorders) | 6 | 3
Stomach Pain (Gastrointestinal disorders) | 2 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 17 | 19
Pancreatic Necrosis (Gastrointestinal disorders) | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Mucositis Oral (Gastrointestinal disorders) | 4 | 1
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 13 | 16
Gastroparesis (Gastrointestinal disorders) | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 1
Lip Pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Esophageal Pain (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2
General Disorders And Administration Site Conditio (General disorders) | 0 | 1
Pain (General disorders) | 9 | 5
Malaise (General disorders) | 3 | 2
Irritability (General disorders) | 1 | 0
Injection Site Reaction (General disorders) | 72 | 68
Flu Like Symptoms (General disorders) | 10 | 9
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Edema Limbs (General disorders) | 3 | 3
Fatigue (General disorders) | 42 | 35
Fever (General disorders) | 17 | 1
Chills (General disorders) | 5 | 2
Infusion Related Reaction (General disorders) | 0 | 1
Allergic Reaction (Immune system disorders) | 4 | 2
Autoimmune Disorder (Immune system disorders) | 1 | 1
Immune System Disorders - Other (Immune system disorders) | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 2 | 1
Skin Infection (Infections and infestations) | 4 | 2
Sinusitis (Infections and infestations) | 2 | 1
Rhinitis Infective (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1
Papulopustular Rash (Infections and infestations) | 1 | 0
Mucosal Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 6
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Bladder Infection (Infections and infestations) | 0 | 1
Injury, Poisoning And Procedural Complications - O (Injury, poisoning and procedural complications) | 0 | 2
Radiation Recall Reaction (Dermatologic) (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Investigations - Other (Investigations) | 3 | 2
Weight Loss (Investigations) | 1 | 1
Weight Gain (Investigations) | 2 | 0
Platelet Count Decreased (Investigations) | 13 | 17
Lymphocyte Count Increased (Investigations) | 0 | 1
Lymphocyte Count Decreased (Investigations) | 4 | 4
Creatinine Increased (Investigations) | 5 | 7
Cholesterol High (Investigations) | 1 | 1
Neutrophil Count Decreased (Investigations) | 16 | 17
Blood Bilirubin Increased (Investigations) | 0 | 1
White Blood Cell Decreased (Investigations) | 18 | 21
Aspartate Aminotransferase Increased (Investigations) | 5 | 6
Alkaline Phosphatase Increased (Investigations) | 7 | 12
Alanine Aminotransferase Increased (Investigations) | 5 | 6
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 7 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 17
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 5
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 6 | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 11 | 10
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 11
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Buttock Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 10
Musculoskeletal And Connective Tissue Disorder - (Musculoskeletal and connective tissue disorders) | 1 | 1
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Nervous System Disorders - Other (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 14 | 19
Peripheral Motor Neuropathy (Nervous system disorders) | 2 | 1
Paresthesia (Nervous system disorders) | 0 | 4
Memory Impairment (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 9 | 13
Sinus Pain (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 8 | 4
Cognitive Disturbance (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 5
Depression (Psychiatric disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 4 | 5
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 1 | 2
Urinary Urgency (Renal and urinary disorders) | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Urinary Tract Pain (Renal and urinary disorders) | 2 | 3
Urinary Frequency (Renal and urinary disorders) | 3 | 9
Proteinuria (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 3 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 5 | 4
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 1 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal Dryness (Reproductive system and breast disorders) | 3 | 1
Pelvic Pain (Reproductive system and breast disorders) | 2 | 1
Breast Pain (Reproductive system and breast disorders) | 1 | 0
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Induration (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
Pain Of Skin (Skin and subcutaneous tissue disorders) | 2 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 7 | 9
Nail Ridging (Skin and subcutaneous tissue disorders) | 0 | 1
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 4 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Lymphedema (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 3
Hot Flashes (Vascular disorders) | 2 | 3
Hematoma (Vascular disorders) | 2 | 0
Flushing (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No